CLINICAL TRIAL: NCT05975775
Title: Study of Postoperative Complications After Laparoscopic Outpatient Radical Prostatectomy in Patients With Localized Prostate Cancer
Brief Title: Outpatient Laparoscopic Radical Prostatectomy
Acronym: LORP
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00622-43
Record Dates: First submitted 2023-07-25; First posted 2023-08-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ambulatory patient cohort: Patients with prostate cancer for whom an ambulatory laparoscopic radical prostatectomy has been validated at a multidisciplinary consultation meeting.
  Interventions: Procedure: Laparoscopic radical prostatectomy

INTERVENTIONS:
Procedure: Laparoscopic radical prostatectomy — Prostate cancer may require laparoscopic radical prostatectomy, a surgical procedure performed under general anaesthetic.

SUMMARY:
The purpose of the study is to evaluate the incidence of surgery-related complications between Day 0 and Day 30.

DETAILED DESCRIPTION:
This is an observational, prospective, open, non-comparative (single arm), bicentric study.

This study is aimed at patients with prostate cancer for whom an ambulatory laparoscopic radical prostatectomy has been validated at a multidisciplinary consultation meeting. The possibility of performing this procedure on an outpatient basis is left to the surgeon's discretion, according to well-defined medical procedure criteria.

This cohort is part of the usual care. The study will observe the incidence and describe the type, number, severity, duration and frequency of procedure-related complications that may arise in the first month post-op of ambulatory Laparoscopic Radical Prostatectomy. For this reason, patient follow-up will stop at 1 month after surgery, during a routine follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male, age ≥ 18 years;
* Localized prostate cancer;
* Validation in a multidisciplinary consultation meeting of curative treatment;
* Scheduled laparoscopic radical prostatectomy;
* Patient able to understand the information related to the study, to read the information leaflet and to signify his/her non-opposition or opposition to participating in the study;
* Membership of a social security scheme;
* Patient having been informed and having given oral non-opposition.

Exclusion Criteria:

* Surgical emergency;
* Patient not eligible for ambulatory care;
* Long-term curative anti-coagulant treatment;
* Resident more than 100km from the clinic;
* Home alone the first night;
* Patient under guardianship, curatorship or deprivation of liberty.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is aimed at patients with prostate cancer for whom an ambulatory laparoscopic radical prostatectomy has been validated at a multidisciplinary consultation meeting. Ambulatory management is at the surgeon's discretion, according to well-defined medical procedure criteria.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | 30 days
  The primary endpoint was the incidence of procedural complications between Day 0 and Day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France